CLINICAL TRIAL: NCT04520672
Title: Circulating Tumor Cells (CTC) in Cancer
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00014; me19Vetter
Record Dates: First submitted 2020-08-05; First posted 2020-08-20 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: circulating tumor cells (CTCs); CTC clusters; Molecular analysis of CTCs; CTC culture; overall survival (OS); progression free survival (PFS)
MeSH Terms: conditions — Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CTC cultures stored in the refrigerator. A "Biobank Reglement" is enclosed to this protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood samples — Blood samples (3 ethylenediaminetetraacetic acid (EDTA) tubes with a volume of 7.5 ml blood each) will be processed for CTC isolation and characterization, ranging from molecular analysis to culture and drug screen.
Other: Samples from tumor draining vessels — In case of tumor resection, 3 EDTA tubes (5 ml) will be withdrawn from the tumor draining vessels for CTC isolation and characterization, ranging from molecular analysis to culture and drug screen.

SUMMARY:
This observational study with circulating tumor cells (CTC) count, isolation and analysis at several time points during disease progression is to investigate the role and biology of CTCs and clusters of CTCs in different cancer types. It also evaluates the role of CTCs as biomarkers, and aims at the identification of key signaling networks that are active in CTCs.

ELIGIBILITY:
Inclusion Criteria:

* Adult cancer patients
* All patients with histology-based proved diagnosis of cancer, all stages and subtypes can be included. Precancerous lesions cannot be included.
* All patients with the diagnosis of a solid tumor including adenocarcinoma, squamous cell carcinoma, neuroendocrine carcinoma, sarcoma
* Written pathology report must be available.
* Written informed consent.

Exclusion Criteria:

* No written informed consent.
* No proved diagnosis of malignancy by pathology report.
* Patients with the diagnosis of blood cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients (> 18 years) with a cancer diagnosis
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in heterogeneous cancer population | Screening (Visit 1) until the date of death (assessed up to 240 months)
  overall survival (OS) in heterogeneous cancer population
Change in total number of isolated CTCs | Through study completion, an average of 20 years
  Change in total number of isolated CTCs

SECONDARY OUTCOMES:
Progression free survival (PFS) | Through study completion, an average of 20 years
  progression free survival (PFS) in the different cancer cohorts with different treatment regimes

OTHER OUTCOMES:
Change in circulating tumor DNA (ctDNA) from blood samples | Through study completion, an average of 20 years
  Change in circulating tumor DNA (ctDNA) from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Vetter, PD Dr. med., Principal Investigator — Kantonsspital Baselland, Liestal
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - Department Oncology, Haematology & Immuntherapy, Kantonsspital Baselland, Liestal